CLINICAL TRIAL: NCT04061772
Title: A Prospective Study of Bortezomib Combined With CHEP Regimen in the Treatment of Primary Peripheral T Cell Lymphoma
Brief Title: A Study of Bortezomib Combined With CHEP in Peripheral T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2019-96
Record Dates: First submitted 2019-08-11; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Bortezomib; CHEP
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Bortezomib; Etoposide; Cyclophosphamide; Epirubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCHEP (Experimental): Bortezomib：1.3mg/m2, intravenous drip, d1,d8, every 3 weeks； Etoposide：100mg/m2,intravenous drip, d1-3, every 3 weeks； Cyclophosphamide：750mg/m2,intravenous drip, d1, every 3 weeks； Pharmorubicin：75mg/m2,intravenous drip, d1,every 3 weeks； Prednisone：100mg,tablet by mouth, d1-5, every 3 weeks.
  Interventions: Drug: Bortezomib; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Pharmorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Bortezomib — Bortezomib injection
Drug: Etoposide — Etoposide injection
Drug: Cyclophosphamide — Cyclophosphamide injection
Drug: Pharmorubicin — Pharmorubicin injection
Drug: Prednisone — Prednisone tablet

SUMMARY:
To evaluate the efficacy and safety of bortezomib combined with CHEP regimen in peripheral T cell lymphoma

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the efficacy and safety of bortezomib combined with CHEP in patients with peripheral T cell lymphoma. Primary end point of this study were objective response rate including complete remission rate and partial remission rate.

ELIGIBILITY:
Inclusion Criteria:

* 1) volunteer to participate in the clinical study: fully understand and know the study, and sign the informed consent in person;Willing to follow and able to complete all test procedures.

  2) age: 18~75 years old (including), male or female. 3) peripheral T cell lymphoma confirmed by histopathology: including peripheral T non-specific type, ALK positive interstitial enlarged cell lymphoma, ALK negative interstitial enlarged cell lymphoma, vascular immune maternal lymphoma, and enteropathy T lymphoma.

  4) no previous chemotherapy, radiotherapy, immunotherapy or other anti-tumor therapy.

  5) the ECOG score is 0-2. 6) there must be at least one evaluable or measurable lesion meeting Lugano 2014 criteria (evaluable lesions: PET/CT examination showed increased uptake of lymph nodes or external nodes (higher than liver) and PET/CT and/or CT characteristics consistent with lymphoma manifestations; Measurable lesions: long diameter >15mm in nodular lesions or long diameter >10mm in external nodules, accompanied by increased FDG uptake).The absence of measurable lesions and increased diffuse FDG uptake in the liver should be excluded.

  7) adequate organ and bone marrow function, no serious hematopoietic dysfunction, abnormal heart, lung, liver, kidney function or immune deficiency (no blood transfusion, granulocyte colony stimulating factor or other relevant medical support was received within 14 days before the use of the study drugs) : A) blood routine: absolute count of neutrophils (ANC) ≥1.5 for 109/L (1500/mm3), platelet ≥75 for 109/L, hemoglobin ≥10 g/dL (for bone marrow involvement, platelet ≥50 for 109/L, ANC ≥1.0 for 109/L, hemoglobin ≥8 g/dL).

B) liver function: serum bilirubin ≤1.5 times the upper limit of normal value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤1.5 times the upper limit of normal value (AST allowed if liver is involved, ALT≤5 times the upper limit of normal value).

C) renal function: the upper limit of serum creatinine ≤1.5 times normal value. D) coagulation function: INR≤1.5 times the upper limit of normal value;PT and APTT≤1.5 upper limit of normal (unless subject is receiving anticoagulant therapy and PT and APTT are within the expected range of anticoagulant therapy at time of screening).

8) in cardiac function examination, left ventricular ejection fraction (LVEF) ≥ 50%.

9) the serum pregnancy test was negative, and effective contraceptive measures were taken from the signing of informed consent until 6 months after the last chemotherapy.

Exclusion Criteria:

* 1) NK/T lymphoma or aggressive natural killer cell leukemia. 2) with hemophagocytic syndrome. 3) primary central nervous system lymphoma or secondary central nervous system involvement.

  4) participating in other clinical studies or the first study drug administration is less than 4 weeks from the end of treatment in the previous clinical study.

  5) other malignancies in the past 5 years, except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the breast and carcinoma in situ of the cervix, which have been treated with radical therapy.

  6) previous anti-tumor therapy, including chemotherapy, immunotherapy, radiotherapy, and biological therapy (tumor vaccines, cytokines, or growth factors that control cancer).

  7) major surgery was performed within 28 days before the study began. 8) a patient with a known history of Human Immunodeficiency Virus infection and/or acquired Immunodeficiency syndrome.

  9) patients with active chronic hepatitis b or active hepatitis c.Screening stage of hepatitis b surface antigen or hepatitis c virus antibody positive patients, must further by hepatitis b virus DNA (no more than 1000 iu/ml) and HCV RNA detection (shall not exceed the method detection limit), in the activity of the ruled out the need for treatment after hepatitis b or hepatitis c infection, before the experiment.Hepatitis b carriers, hepatitis b patients who are stable after drug treatment and hepatitis c patients who have been cured can be enrolled.

  10) active tuberculosis. 11) any active infections, including but not limited to bacterial, fungal or viral infections, that require systematic anti-infective therapy within 14 days prior to the initiation of the study.

  12) pregnant or lactating women. 13) patients with uncontrolled concomitant diseases, including but not limited to symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, active peptic ulcer or hemorrhagic diseases.

  14) having a history of mental illness;Having no capacity or limited capacity. 15) the underlying condition of the patient may increase the risk of receiving the study drug, or may cause confusion as to the toxicity and its judgment.

  16) patients considered unsuitable to participate in this study by other researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-08-12 (Estimated); Primary Completion 2021-07-05 (Estimated); Study Completion 2021-12-05 (Estimated)

PRIMARY OUTCOMES:
response rate | up to 18 weeks
  overall response rate including complete response and partial response

SECONDARY OUTCOMES:
adverse effects | through study completion, an average of 30 days
  adverse effects and serious adverse effects
survival outcome | through study completion, at least 1 year
  Progression Free Survival
survival outcome | through study completion, at least 1 year
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chen, PhD, Study Director — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The parimary and secondary end point of the study, the characteristics of patients are to be shared.
Supporting Information: Study Protocol, SAP
Time Frame: after the republication of the main article and for 6 months